CLINICAL TRIAL: NCT04700111
Title: Lag of Accommodation With DOT Spectacle Lenses
Acronym: ASH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2011-001
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myopia, Myopia Progression, Lag of Accommodation, Hyperopic Retinal Blur, Reduction in Contrast
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment 1 - DOT Pattern (Experimental): Spectacle lens or treatment 1
  Interventions: Device: DOT Pattern
- Treatment 2 - Control Spectacles (Active Comparator): Comparator lens or control arm
  Interventions: Device: Control Spectacles

INTERVENTIONS:
Device: DOT Pattern — DOT Pattern Spectacle Lens
  Arms: Treatment 1 - DOT Pattern
Device: Control Spectacles — Control lens
  Arms: Treatment 2 - Control Spectacles

SUMMARY:
The objective of the study is to measure the difference in the lag of accommodation between DOT spectacle lenses and control spectacles.

ELIGIBILITY:
A person is eligible for inclusion in the study if he/she:

1. Age 6-18 years of age, with a maximum of 6 of the first 25 completed participants being older than 14 years of age.
2. Is able to read (or be read to), understand and sign the assent document if under 17 years old or is able to read, understand and sign the consent document if aged 17 or 18 years.
3. Is under 17 years old and is accompanied by a parent or legal guardian who is able to read, understand and sign the parental information and permission document.
4. Should be emmetropic by non-cycloplegic auto-refraction, which means both refractive meridians should be within +1.00D and -1.00D.
5. Is willing and able to follow instructions.

A person will be excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study.
2. Have a history of myopia control treatment in the past year.
3. Has amblyopia in either eye or known to have any other binocular vision disorder, such as accommodative insufficiency.
4. Has any known active ocular disease and/or infection.
5. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable. Examples include diabetes mellitus, hyperthyroidism.
6. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable. Examples include Atropine eye drops.
7. Has undergone strabismus surgery, refractive error surgery or intraocular surgery.
8. Is a child of a member of the study team.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Best vision sphere | 90 minutes
  1) Autorefractor spherical equivalent refraction measured at distance and at 40cm with each pair of treatment spectacles

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research and Education, Waterloo, Ontario, Canada